CLINICAL TRIAL: NCT05727683
Title: A Phase I Open, Single-arm Study of JWCAR029 (CD19-targeted Chimeric Antigen Receptor T Cells) for Patients With Relapsed or Refractory in B-cell Acute Lymphoblastic Leukemia
Brief Title: CD19-targeted CAR T Cells for Patients With Relapsed or Refractory in B-cell Acute Lymphoblastic Leukemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Ming Ju Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JWCAR029-006
Record Dates: First submitted 2023-02-05; First posted 2023-02-14 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Acute Lymphocytic Leukemia
Keywords: JWCAR029; Relapsed/Refractory; Pediatric and young adults
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Recurrence | interventions — Automobiles; fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JWCAR029 Treatment (Experimental): A lymphodepletion conditioning with cyclophosphamide and fludarabine will be conducted before JWCAR029 infusion.
  Potential JWCAR029 doses:
  Dose level 1: 0.10×10^6 CAR+ T cells/kg Dose level 2: 0.30×10^6 CAR+ T cells/kg Dose level 3: 0.75×10^6 CAR+ T cells/kg Dose level 4: 1.0×10^6 CAR+ T cells/kg
  Interventions: Biological: CD19-targeted Chimeric Antigen Receptor (CAR) T Cells

INTERVENTIONS:
Biological: CD19-targeted Chimeric Antigen Receptor (CAR) T Cells — Subjects will receive Lymphodepleting chemotherapy with intravenous (IV) fludarabine (25 mg/m2/day for 3 days) plus cyclophosphamide IV (250 mg/m2/day for 3 days) (flu/cy) concurrently, followed by JWCAR029 cells infusion. Phase 1 will evaluate up to 4 JWCAR029 cells dose levels.
  Other Names: Fludarabine; Cyclophosphamide

SUMMARY:
This is a phase I, open-label, single-arm study conducted in China to evaluate the safety, tolerability, PK, and determine the recommended phase II dose (RP2D) and/or maximum tolerated dose (MTD) (if applicable) of JWCAR029 in pediatric and young adult subjects with r/r B-ALL.

DETAILED DESCRIPTION:
Dose exploration for this study will be a 3+3 design with a target DLT rate of <1/3. Dose exploration can be discontinued once one or more dose levels with an acceptable safety profile and satisfactory antitumor activity have been selected for subsequent evaluation. The maximum tolerated dose (MTD) may not be achieved at the dose levels predetermined in this study as described below.

During the treatment period of the study, four dose levels of JWCAR029 will be evaluated. enrollment will begin at dose level 1, follow a 3+3 dose exploration design protocol, and finally select one or more dose levels with an acceptable safety profile and good antitumor activity as the recommended dose, after which dose exploration will be discontinued.

Dose limiting toxicity (DLT) will be evaluated within 28 days after JWCAR029 infusion. Each dose cohort is planned to enroll three subjects initially, and at least one pediatric subject younger than 10 years of age who can be evaluated for DLT will be enrolled at each dose level. In the first dose cohort, the first 3 subjects will be infused at least 14 days apart. At each higher dose level, the first 3 patients within the dose cohort will be treated at least 7 days apart. For dose levels considered safe, at least 3 subjects with assessable DLT must complete a 28-day DLT assessment period.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≤ 30 years and weight ≥10kg.
2. Patients with r/r B-ALL, defined as morphological disease in the bone marrow(≥5% blasts) and either of the following:

   * ≥2 BM relapse;
   * Refractory defined as relapse if first remission<12 months or not achieving a CR after 1 cycle of a standard induction chemotherapy regimen for relapsed leukemia;primary chemo-refractory as defined by not achieving a CR after 1 cycle of a conventional chemotherapy or 2 cycles of a standard induction chemotherapy regimen for relapsed leukemia;
   * Any BM relapse after HSCT which must be ≥90 days from HSCT at the time of screening, and be required free from GVHD and ended from any immunosuppressive therapy ≥1 month at the time of screening;
   * Patients with Ph+ ALL are eligible if they are intolerant to or have failed two lines of TKI therapy, or if TKI therapy is contraindicated.

   Note: Patients with MRD+ after bridging therapy will be allowed for treatment.
3. Karnofsky (age ≥16 years) or Lansky (age <16 years) performance status >60.
4. Adequate organ function.
5. Vascular access is sufficient for leukocyte isolation.
6. Expected survival time > 3 months.
7. Any non-hematological toxicity due to previous treatment, except for alopecia and peripheral neuropathy, must be restored to ≤ grade 1.
8. Females of childbearing potential (all female subjects who are physiologically capable of becoming pregnant) must agree to use a highly effective method of contraception for 1 year following JWCAR029 infusion; male subjects whose partners are of childbearing potential must agree to use an effective barrier method of contraception for 1 year following JWCAR029 infusion.

Exclusion Criteria:

1. leukemic CNS involvement with active CNS lesions and significant neurodegenerative manifestations, or subjects with CNS grade CNS-2/CNS-3 as assessed by NCCN guidelines (subjects rated CNS-2 due to puncture injury may be enrolled).
2. existing or previous clinically significant CNS lesions such as epilepsy, epileptic seizures, paralysis, aphasia, cerebral edema, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, psychosis, etc.
3. Patients with genetic syndromes other than Down syndrome.
4. Patients with Burkitt's lymphoma.
5. History of malignancy other than B-ALL for at least 2 years prior to enrollment.
6. Subject has HBV, HCV, HIV or syphilis infection at the time of screening.
7. Subject has deep vein thrombosis (DVT) (cancer thrombosis or thrombosis) or pulmonary artery embolism (PE) or is on anticoagulation therapy for DVT or PE within 3 months prior to signing the informed consent form
8. uncontrolled systemic fungal, bacterial, viral or other infections.
9. Combination of active autoimmune diseases requiring immunosuppressive therapy.
10. Acute or chronic graft-versus-host disease.
11. History of any of the following cardiovascular diseases within the past 6 months: Class III or IV heart failure as defined by the New York Heart Association (NYHA), cardiac angioplasty or stenting, myocardial infarction, unstable angina, or other clinically significant heart disease.
12. Women who are pregnant or lactating. Women of childbearing potential must have a negative serum pregnancy test within 48 hours prior to initiation of lymphocyte clearance chemotherapy.
13. Previous treatment with CAR-T cells or other gene-modified T cells.
14. Previous anti-CD19/anti-CD3 therapy, or any other anti-CD19 therapy.
15. Relevant medications or treatments within a specified time frame.
16. The presence of any factors affecting the subject's compliance with the protocol, including uncontrollable medical, psychological, family, sociological, or geographic conditions, as determined by the investigator; or unwillingness or inability to comply with the procedures required in the study protocol.
17. Known life-threatening allergic reactions, hypersensitivity reactions, or intolerance to JWCAR029 cell formulation or its excipients.

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Estimated)
Dates: Start 2022-04-28 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Experiencing Dose Limiting Toxicities (DLTs) | Day 28 after JWCAR029 infusion
  Dose limiting toxicity (DLT) is an AE that meets the following criteria and occurs within 28 days of JWCAR029 infusion.AE is graded according to CTCAE version 5.0, CRS is graded according to the American Society for Transplantation and Cellular Therapy (ASTCT) 2019 consensus CRS grading criteria, and neurotoxicity is graded according to the ASTCT 2019 consensus ICANS grading criteria.
The occurrence of adverse events | After JWCAR029 infusion for 2 year
  These adverse events would be measured by assessment scale method according to NCI CTC AE v5.0 classification standard

SECONDARY OUTCOMES:
Overall remission Rate | After JWCAR029 infusion for 2 year
  Overall remission rates assessed by investigators at 1, 2, and 3 months after JWCAR029 infusion,Include complete remission (CR) and complete morphological remission without complete recovery of blood counts （CRi），and the results of the efficacy assessment at each time point
MRD negative rate | After JWCAR029 infusion for 2 year
  Investigator assessed response rate for microscopic residual disease (MRD) at 1 , 2 and 3 months after completion of infusion, including the percentage of patients achieving MRD negativity (MRD level <10^-4) among all infused patients

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofan Zhu, PhD, Principal Investigator — Hematology Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Hematology Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No